CLINICAL TRIAL: NCT00511901
Title: Prevalence and Treatment of Anemia in Patients Admitted to Subacute Rehabilitation Hospital
Brief Title: Prevalence and Treatment of Anemia in Rehabilitation Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study enrollment was suspended in response to an FDA alert regarding the study drug. The study was subsequently terminated
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220045106
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2011-11

CONDITIONS: Anemia
Keywords: anemia; function; rehabilitation
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; Niferex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo & Niferex (Placebo Comparator): Placebo (for epoetin alpha) subcutaneous injection weekly for 8 weeks and Niferex 150 mg twice a day for 8 weeks
  Interventions: Drug: placebo; Drug: Niferex
- epoetin alpha & Niferex (Active Comparator): 40,000 IU (initial dose) epoetin alpha subcutaneous injection weekly for 8 weeks and Niferex 150 mg twice a day for 8 weeks
  Interventions: Drug: epoetin alpha; Drug: Niferex

INTERVENTIONS:
Drug: placebo
  Arms: Placebo & Niferex
Drug: epoetin alpha
  Other Names: Procrit
  Arms: epoetin alpha & Niferex
Drug: Niferex
  Other Names: iron polysaccharide

SUMMARY:
Patients who are admitted to subacute rehabilitation facilities following hospitalization are frequently anemic. The purpose of this study is to see if anemic patients treated with epoetin alfa will have higher hemoglobin levels and better functional recovery at 3, 8, and 12 weeks after study entry compared to patients who do not receive epoetin alfa.

DETAILED DESCRIPTION:
Anemia is associated with loss of function in some studies. However, it is unknown if more rapid correction of anemia in patients who enter a rehabilitation setting after surgery or from hospitalization for acute medical problems leads to shorter rehabilitation stays and improved functional status.

Patients aged 60 and older who have hemoglobin levels of less than 10.5 g/dL will be randomized to receive 8 weekly doses of either erythropoietin alfa or placebo. Functional status will be measured at baseline and then at 3, 8 and 12 weeks.

The following specific aims will be tested in this study:

* Determine the prevalence of anemia in patients admitted to a subacute rehabilitation facility with potential for recovery.
* Determine the baseline functional status of patients admitted to a subacute rehabilitation facility with potential for recovery using the Functional Independence Measure (FIM), an assessment tool used in acute rehabilitation settings.
* Determine if administration of epoetin alfa will result in higher hemoglobin concentrations in patients receiving the drug than in patients given placebo at 3, 8 and 12 weeks after entry into the study.
* Perform a study that establishes the feasibility of a trial to test whether epoetin alfa produces improvements in the FIM, grip strength, the time it takes for patients to reach rehabilitation goals, activity monitor, fatigue, mood, functional recovery and reduces length of rehabilitation stay.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Admission hemoglobin concentration of < 10.5 g/dL.
* Able to read and understand English.
* Consent signed by subjects.

Exclusion Criteria:

* Unable to randomize within 7 days of admission to rehabilitation center.
* Folstein min-mental status score of < 21.
* Neuromuscular disease and/or disability; in clinical judgment of the investigators that do not have rehabilitation potential.
* Diagnosis or evidence of carcinoma (excluding skin cancer other than melanoma) within the past five years
* Admission for stroke with residual deficit
* Wheelchair bound prior to acute event.
* Dialysis dependent chronic renal failure
* Home more than 1 hour drive from hospital.
* Admitted to long term nursing or hospice care.
* Active blood loss.
* Known history of severe iron deficiency.
* Hematological disease that results in anemia that may not respond to erythropoietin (including, but not limited to, myelodysplastic syndrome, hematological malignancy, hemolytic syndromes, hemoglobinopathy).
* Uncontrolled hypertension (systolic BP >200 mmHg or diastolic BP >110 mmHg) after adequate antihypertensive therapy.
* New onset seizures (within three months) or seizures not controlled by medication.
* Objective diagnosis of pulmonary embolism or deep vein thrombosis within the past 10 years.
* Patients with a condition (e.g. psychiatric illness) or in a situation that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's compliance with study procedures.
* Acute burns.
* Treatment with any recombinant human erythropoietin within 30 days prior to enrollment.
* Known hypersensitivity to human albumin or mammalian cell-derived products or recombinant human erythropoietin (rHuEPO).
* Received an experimental drug or used an experimental medical device within 30 days prior to the planned start of treatment.
* Pregnancy or lactation.
* Employees of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Elms of Cranbury, Cranbury, New Jersey
  - Care One East Brunswick, East Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited at two subacute rehabilitation facilities in Central New Jersey between October 2005 and March 2008
Period: Overall Study
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Started | 11 | 11
Completed | 10 | 8
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intention to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (8.3) | 75.5 (8.4) | 75.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 9 | 10 | 19
  Black | 2 | 1 | 3
Hemoglobin Level [Mean (Standard Deviation); unit: g/dL] — Level Prior to Randomization
  g/dL | 9.8 (1.0) | 9.8 (0.6) | 9.8 (0.8)
Days From Admit to Randomization [Mean (Standard Deviation); unit: Days] — # of days from admission to the subacute rehabilitation facility to randomization into the study
  Days | 5.5 (1.5) | 5.3 (1.8) | 5.4 (1.6)
FIM Motor Scale [Mean (Standard Deviation); unit: Scores on a Scale] — The Functional Independence Measure scale is a 7 point rating scale used as part of the Uniform Data System for Medical Rehabilitation. The FIM motor score ranges from 13 to 91 (most independent).
  Scores on a Scale | 74.2 (8.8) | 68.8 (6.9) | 71.5 (8.2)
FACIT Fatigue Scale [Mean (Standard Deviation); unit: Scores on a Scale] — FACIT-Fatigue Scale (version 4) 13 item questionnaire to assess level of fatigue. The FACIT-Fatigue scores range from 0 to 52(most fatigue).
  Scores on a Scale | 31.6 (9.5) | 29.2 (11.6) | 30.4 (10.4)
POMS Depression-Dejection Scale [Median (Inter-Quartile Range); unit: Scores on a Scale] — Profile of Mood States (POMS) Depression-Dejection Scale 15 item questionnaire to measure the degree of depressive thoughts. The POMS scores range from 0 to 60(most depressed).
  Scores on a Scale | 3 [1 to 13] | 3 [0 to 8] | 3 [1 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Mean Hemoglobin Concentration at 8 Weeks After Entry Into the Study
Time Frame: 8 weeks following randomization
Population: Intention to treat; of the subjects not lost to follow-up, 3 subjects in the placebo arm & 2 subjects in the epoetin alpha arm were not available for 8 week hemoglobin draw
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 7 | 6
g/dL | 11.9 (1.2) | 13.6 (0.6)
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.7

2. Secondary Outcome: Motor-FIM Score
Description: FIM Motor score ranges from 13 to 91 (most independent)
Time Frame: 3, 8, and 12 weeks following randomization
Population: exact numbers of subjects analyzed at each time point vary based on time of study withdrawal for those who withdrew and availability of subject for those who were under active follow-up
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 10 | 9
Scores on a Scale
  FIM at 3 weeks (n=9; n=9) | 76.9 (4.4) | 77.7 (5.7)
  FIM at 8 weeks (n=9; n=7) | 81.7 (4.2) | 85.0 (4.4)
  FIM at 12 weeks (n=10; n=8) | 85.2 (3.8) | 85.1 (5.8)
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; FIM at 3 weeks; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Mean Difference (Net) = .8
Statistical Analysis 2: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; FIM at 8 weeks; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 3.3
Statistical Analysis 3: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; FIM at 12 weeks; Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.1

3. Secondary Outcome: Length of Stay in Subacute Rehabilitation Facility
Description: Days from randomization to discharge
Time Frame: 12 weeks following randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 10 | 11
Days | 13.1 (5.2) | 17.4 (9.0)
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 4.3

4. Secondary Outcome: Grip Strength
Description: kilograms measured by hand held dynamometer
Time Frame: 3, 8, and 12 weeks following randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 10 | 10
kg
  Grip Strength at 3 weeks (n=9; n=10) | 19.0 (4.0) | 18.4 (3.1)
  Grip Strength at 8 weeks (n=9; n=7) | 19.4 (3.7) | 19.6 (4.2)
  Grip Strength at 12 weeks (n=10; n=8) | 17.4 (3.5) | 19.0 (3.6)
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Grip strength at 3 weeks; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.6
Statistical Analysis 2: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Grip strength at 8 weeks; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.2
Statistical Analysis 3: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Grip strength at 12 weeks; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.6

5. Secondary Outcome: Short Physical Performance Battery (SPPB) Score
Description: Measure physical function scored 0 - 12 (better)
Time Frame: 3, 8, and 12 weeks following randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 10 | 9
Scores on a scale
  SPPB at 3 weeks (n=9; n=9) | 3.4 (1.9) | 3.7 (2.5)
  SPPB at 8 weeks (n=9; n=7) | 7.0 (1.9) | 7.4 (2.9)
  SPPB at 12 weeks (n=10; n=8) | 8.0 (2.3) | 7.1 (3.1)
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; SPPB at 3 weeks; Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.3
Statistical Analysis 2: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; SPPB at 8 weeks; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.4
Statistical Analysis 3: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; SPPB at 12 weeks; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.9

6. Secondary Outcome: FACIT Measurement System Fatigue Scale
Description: Fatigue score ranges from 0 to 72. Lower score represents less fatigue
Time Frame: 3, 8, and 12 weeks following randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 10 | 9
Scores on a Scale
  FACIT at 3 weeks (n=8; n=9) | 38.3 (6.7) | 35.7 (10.7)
  FACIT at 8 weeks (n=9; n=7) | 39.8 (11.2) | 42.3 (8.3)
  FACIT at 12 weeks (n=10; n=8) | 42.7 (6.7) | 38.6 (10.4)
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; FACIT at 3 weeks; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -2.6
Statistical Analysis 2: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; FACIT at 8 weeks; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.5
Statistical Analysis 3: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; FACIT at 12 weeks; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -4.1

7. Secondary Outcome: Activity Counts
Description: Activity counts as measured by the Actigraph monitor. Higher counts indicate more activity.
Time Frame: 3, 8, and 12 weeks following randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 10 | 9
Counts
  Activity Counts at 3 weeks (n=8; n=9) | 51.13 (27.0) | 41.56 (28.1)
  Activity Counts at 8 weeks (n=9; n=6) | 58.78 (32.8) | 70.17 (27.3)
  Activity Counts at 12 weeks (n=10; n=8) | 61.60 (27.2) | 77.75 (44.6)
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Activity Counts at 3 weeks; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -9.57
Statistical Analysis 2: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Activity Counts at 8 weeks; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 11.39
Statistical Analysis 3: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; Activity Counts at 12 weeks; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 16.15

8. Secondary Outcome: POMS Depression-Dejection Scale
Description: Profile of Mood States (POMS) Depression-Dejection Scale 15 item questionnaire to measure the degree of depressive thoughts. The scale ranges from 0 to 60 (most depressed).
Time Frame: 3,8,12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Scores on a Scale
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Number analyzed (Participants) | 10 | 10
Scores on a Scale
  POMS at 3 weeks (n=9; n=10) | 1 [0 to 7] | 3.5 [0 to 8]
  POMS at 8 weeks (n=9; n=7) | 1 [0 to 5] | 0 [0 to 8]
  POMS at 12 weeks (n=10; n=7) | 1 [0 to 2] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; POMS at 3 weeks; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney); Median Difference (Net) = 2.5
Statistical Analysis 2: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; POMS at 8 weeks; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1
Statistical Analysis 3: Comparison: Placebo & Niferex vs Epoetin Alpha & Niferex; POMS at 12 weeks; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: active followup at 3, 8, & 12 weeks
Arm/Group | Placebo & Niferex | Epoetin Alpha & Niferex
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo & Niferex (N=11) | Epoetin Alpha & Niferex (N=11)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Hip Fracture

LIMITATIONS AND CAVEATS:
Limited number of eligible subjects, burdensome protocol requirements impeded recruitment, controversy concerning safety of epoetin alpha which led to early termination of study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes